CLINICAL TRIAL: NCT00496236
Title: A Phase I/II Safety, Tolerability and "Proof of Concept" Study of Radiotherapy, Cetuximab, and Intratumoral Injections of TNFerade™ Biologic (AdGVEGR.TNF.11D) for Elderly or Frail Patients or Intermediate Stage Patients With Head and Neck Cancer
Brief Title: Radiotherapy, Cetuximab, and Injections of TNFerade™ Biologic for Elderly or Frail Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GenVec (Industry)
Responsible Party: Paul Fischer, PhD, GenVec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GV-001.010; GV-001.010 (TNF-ELF)
Record Dates: First submitted 2007-06-28; First posted 2007-07-04 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2011-05

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms
Keywords: head; neck; cancer; neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

INTERVENTIONS:
Drug: TNFerade biologic

SUMMARY:
This study is looking at the safety and tolerability of TNFeradeä Biologic combined with conventional once daily radiation therapy in elderly or frail patients with new onset locally advanced head and neck tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or older with an ECOG performance status 0-2,or
* Patients > 18 years of age with ECOG performance status of 2 or greater, or
* Patients > 18 years of age unsuitable for concurrent chemotherapy or surgery due to:
* Renal failure, or
* Severe cardiopulmonary disease, or
* Other end-organ dysfunction that precludes the use of chemotherapy but does not preclude the administration of TNFerade™ Biologic or cetuximab
* Tumor that is unresectable or inoperable and not amenable to regular concurrent chemoradiotherapy
* Patients > 18 years of age with intermediate stage disease, stages II-III (T2-T3, N0-1MO) carcinoma of the head and neck, including oral cavity, pharynx larynx, paranasal sinuses and cervical esophagus. Selected patients with stage IV disease (T4N0-1M0) will also be considered for enrollment. Therapy is given with curative intent.
* Disease should be clinically accessible (measurable or evaluable) to keep injection via direct intratumoral injection
* Informed consent

Exclusion Criteria:

* History of malignancy in the last 2 years except carcinoma in situ of the cervix or bladder, non-melanomatous skin cancer, or localized early stage prostate cancer, with patients continually disease free, or cancers that are not felt to influence treatment for head and neck cancer and life expectancy of patient
* Overt systemic metastatic disease
* Previous radiation or chemotherapy for malignancy of the head and neck
* Clinical evidence of active infection of any type
* pregnant or lactating women
* Experimental medications within the last 4 weeks prior to Day 1
* Chronic treatment for greater than 6 months with steroids at doses above 10 mg/day prednisone (or equivalent)
* Patients receiving hormone replacement therapy or hormonal contraceptives within 2 weeks of day 1
* Patients who have undergone surgery within the last 1 month
* Allergic reaction to cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
The maximum tolerated dose established in the Phase I (dose-finding) portion of the study will be used to assess the investigational drug's ability to enhance clinical outcome. The primary endpoint being locoregional control rate at 24 months.

SECONDARY OUTCOMES:
Locoregional control at 3,6, and 12 months, objective response rate, progression-free survival at 3,6,12, and 24 months, and the rate of distal metastases at 3,6, 12 and 24 months will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes,, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States